CLINICAL TRIAL: NCT04306120
Title: Neurorehabilitation Lab at Department of Physical Therapy in KMU
Brief Title: Effects of Thermal Stimulation on Motor Recovery and Neuromuscular Property of Lower Extremity in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, KMUHIRB-F(II)-20200009, Principal Investigator, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20200009
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Cardiovascular
Keywords: Thermal stimulation; Stroke; Spinal circuit; Motor function; Lower extremity
MeSH Terms: conditions — Myocardial Infarction; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- noxious cold group (Active Comparator): The group received noxious cold (3 - 4°C) stimuli on the affected leg for 30 minutes.
  Interventions: Other: Traditional Rehabilitation Therapy
- noxious heat group (Active Comparator): The group received noxious heat (46 - 47°C) stimuli on the affected leg for 30 minutes.
  Interventions: Other: Traditional Rehabilitation Therapy
- alternative thermal stimulation group (Active Comparator): The group received alternative noxious heat (46 - 47°C) and noxious cold (3 - 4°C) stimuli on the affected leg for 30 minutes.
  Interventions: Other: Traditional Rehabilitation Therapy

INTERVENTIONS:
Other: Traditional Rehabilitation Therapy — The protocol included range of motion, ambulation, endurance, strengthening, reconditioning exercise, and home program education according to therapists' plans and the patients' ability.

SUMMARY:
This 3-year study will recruit a total of 72 subjects with first-ever stroke after 3 months onset from the department of Physical Medicine and Rehabilitation in 3 teaching hospitals. This study design employs a prospective single-blinded, randomized controlled trial with pretest, posttest, and follow-up assessments. Participants who meet and be willing to join this study will be assigned into one of three groups (noxious cold only, noxious heat only, or alternative TS). All subjects will receive conventional rehabilitation. In addition, three groups will receive an additional TS protocol with a total of 15 sessions for 3 weeks (5 times per week, 30 minutes daily). Primary outcome measures include the LE subscale of Fugl-Meyer assessment, the modified Ashworth scale, the Postural Assessment Scale for Stroke Patients, Timed Up and Go test, and the Barthel index. Moreover, spinal circuit excitability will be assessed by measuring Hoffmann reflex/ M wave ratio, H-reflex recruitment curves, and reciprocal inhibition of the soleus muscle. Muscle properties will be evaluated by measuring the soleus muscle tone, elasticity, and stiffness. All participants will be assessed with the outcome measures at beginning of the intervention, the end of the intervention, 1 month and 3 months after the intervention.

DETAILED DESCRIPTION:
Effective evaluation and treatment for lower extremity (LE) motor and function recovery in patients with stroke have been one of the primary goals for rehabilitation therapy. The purposes of this study are to compare immediate and long-term treatment effects among noxious cold only, noxious heat only, and alternative thermal stimulation (TS) on the LE motor recovery and neuromuscular properties and to investigate the relationships among spinal circuit excitability, muscle properties, and motor function of LE in patients with chronic stroke.

This 3-year study will recruit a total of 72 subjects with first-ever stroke after 3 months onset from the department of Physical Medicine and Rehabilitation in 3 teaching hospitals. This study design employs a prospective single-blinded, randomized controlled trial with pretest, posttest, and follow-up assessments. Participants who meet and be willing to join this study will be assigned into one of three groups (noxious cold only, noxious heat only, or alternative TS). All subjects will receive conventional rehabilitation. In addition, three groups will receive an additional TS protocol with a total of 15 sessions for 3 weeks (5 times per week, 30 minutes daily). Primary outcome measures include the LE subscale of Fugl-Meyer assessment, the modified Ashworth scale, the Postural Assessment Scale for Stroke Patients, Timed Up and Go test, and the Barthel index. Moreover, spinal circuit excitability will be assessed by measuring Hoffmann reflex/ M wave ratio, H-reflex recruitment curves, and reciprocal inhibition of the soleus muscle. Muscle properties will be evaluated by measuring the soleus muscle tone, elasticity, and stiffness. All participants will be assessed with the outcome measures at one week before the intervention, beginning of the intervention, the end of the intervention, 1 month and 3 months after the intervention. A two-way repeated measures analysis of variance will be used to investigate the effects among the three groups across time points tested with adequate post-hoc comparisons.

The results of this study will help to understand the immediate and long-term effects of motor recovery of different TS modes and the adaptive change of neuromuscular properties as well to select the more effective TS treatment mode on facilitating LE motor and function recovery in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate to this study with written informed consent
2. First-ever stroke
3. More six months after stroke onset
4. Ability to maintain an independent sitting posture for at least 30 minutes
5. Mini Mental Status Examination score more than 24

Exclusion Criteria:

1. Skin disease, skin injuries, burns, or fresh scars over the thermal stimulation application area
2. Contraindication of ice or heat application
3. Uncontrolled blood pressure and heart conditions
4. History of diabetes with known peripheral vascular pathology
5. Pregnancy
6. Unable to communicate with simple instruction or aphasia
7. Receiving Botulinum toxin drug treatment
8. Considered as unsuitable by the principal investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
The Lower Extremity subscale of Fugl-Meyer assessment (FMA-LE) | Change from the beginning of the intervention to the end of the intervention, 1 month and 3 months after the intervention.
  The FMA-LE consists of 17 items, each scored on a 3-point scale (0 to 2). The total score of the FMA-LE ranges from 0 to 34, and higher scores indicate better motor performance.
The Postural Assessment Scale for Stroke (PASS) | Change from the beginning of the intervention to the end of the intervention, 1 month and 3 months after the intervention.
  The PASS is a 4-point rating (0 to 3) scale with well-established reliability and validity that measures balance function in persons with stroke. The total score of the PASS ranges from 0 to 36, and higher scores indicate greater balance function.
The modified Ashworth scale (MAS) | Change from the beginning of the intervention to the end of the intervention, 1 month and 3 months after the intervention.
  The modified Ashworth scale is a 6-point rating scale (0 to 5) with well-established inter-rater reliability that measures muscle tone of ankle plantarflexor in persons with stroke. Higher MAS scores indicate greater severity of spasticity.
The Barthel index (BI) | Change from the beginning of the intervention to the end of the intervention, 1 month and 3 months after the intervention.
  The Barthel index is used to evaluate activity of daily living function.The Barthel index consists of 10 items. The total score of the Barthel index ranges from 0 to 20, and higher scores indicate better outcome.
Timed up and go test(TUG) | Change from the beginning of the intervention to the end of the intervention, 1 month and 3 months after the intervention.
  The Timed Up and Go (TUG) test assesses mobility by measuring the time it takes for someone to stand, walk a short distance, turn, and sit back down. Faster times suggest better mobility, while longer times may indicate mobility limitations or fall risk. It's a useful tool to evaluate functional capacity and guide interventions for improved mobility.

SECONDARY OUTCOMES:
Spinal circuit excitability | Change from the beginning of the intervention to the end of the intervention, 1 month and 3 months after the intervention.
  Spinal circuit excitability will be assessed by measuring Hoffmann reflex/ M wave ratio of the soleus muscle. Higher scores indicate poorer outcome.
Muscle properties | Change from the beginning of the intervention to the end of the intervention, 1 month and 3 months after the intervention.
  Muscle properties will be evaluated by measuring the soleus muscle stiffness. Higher scores indicate poorer outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Hong Lin, PhD, Principal Investigator — Department of Physical Therapy
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Select One..., Taiwan

IPD SHARING:
Plan to Share IPD: No